CLINICAL TRIAL: NCT06522334
Title: Interstitial Lung Disease Registry Study: Prospective and Retrospective Observational Study in Austria
Status: Recruiting | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Lung Health (Other)
Responsible Party: Principal Investigator, Robab Breyer-Kohansal, Head of Department for Internal Medicine and Pneumology Clinic Hietzing, Ludwig Boltzmann Institute for Lung Health
Other Study IDs: ILD Registry
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this registry is to systematically record epidemiological and clinical data throughout the whole interstitial lung disease course - starting with the diagnosis, therapy, follow up of lung function, symptom control, adverse events, medication, survival and death.

There are no additional interventions regarding this registry.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of interstitial lung disease
* written informed consent

Exclusion Criteria:

* to not comprehend and rightfully judge participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Everybody with a diagnosis of interstitial lung disease, over 18 years old will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2034-02-28 (Estimated); Study Completion 2034-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 years
  Mortality caused by interstitial lung disease
Loss of lung function | 2 years
  FVC and DLCO loss within 24 months

SECONDARY OUTCOMES:
Prevalence | 10 years
  Prevalence of the different interstitial lung diseases in Austria
Response to drugs | 10 years
  Response to immunosuppressive/immunomodulating/antifibrotic drugs

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (5):
  - Klinik Hietzing, Vienna
  - Klinik Penzing, Vienna
  - Ludwig Boltzmann Institut for Lung Health, Vienna
  - Klinik Ottakring, Vienna
  - Klinik Floridsdorf, Vienna